CLINICAL TRIAL: NCT01916148
Title: Expanded Access Use of 18F-L-Fluoro-DOPA PET/CT Scan Localization of Focal Pancreatic Lesions in Subjects With Hyperinsulinemic Hypoglycemia
Brief Title: 18F-L-Fluoro-DOPA PET/CT Scan Localization of Focal Pancreatic Lesions in Subjects With Hyperinsulinemic Hypoglycemia
Status: Available | Type: Expanded Access
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Lisa States, Principal Investigator, Children's Hospital of Philadelphia
Other Study IDs: 12-009528
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Congenital Hyperinsulinism (CHI); Beckwith-Wiedemann Syndrome; Insulinoma
Keywords: Hypoglycemia; Hyperinsulinism (HI); F-DOPA; PET; 18-F DOPA; 18F-L-Fluoro-DOPA; 18F-fluoro-L-dihydroxyphenylalanine; focal pancreatic lesions; congenital hyperinsulinism; Beckwith Wiedemann Syndrome; insulinoma; Hyperinsulinemic Hypoglycemia; F-DOPA PET; CHI (Congenital hyperinsulinism)
MeSH Terms: conditions — Congenital Hyperinsulinism; Beckwith-Wiedemann Syndrome; Insulinoma; Hypoglycemia; Hyperinsulinism | interventions — fluorodopa F 18

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: 18F-DOPA — 18F-DOPA is a PET (Positron Emission Tomography) scan radiotracer.
  Other Names: 18F-fluoro-L-dihydroxyphenylalanine; 18F-L-Fluoro-DOPA

SUMMARY:
This purpose of this study is to determine the ability of an 18F-fluoro-L-dihydroxyphenylalanine (18F-DOPA) PET (Positron Emission Tomography) scan to detect a focal lesion of hyperinsulinism and determine the location in patients with congenital hyperinsulinism, Beckwith Wiedemann Syndrome and suspected insulinoma. Safety data will be collected.

DETAILED DESCRIPTION:
Patients with hyperinsulinemic hypoglycemia are at risk for neurological damage due to hypoglycemia. Early surgical intervention can be preventative. F-DOPA PET may be able to detect of a focal lesion prior to surgical intervention and be used during surgical planning to guide the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any age with hyperinsulinemic hypoglycemia, diagnosed by a fasting test and/or response to glucagon stimulation.
* Subjects who are eligible for pancreatic surgery regardless of prior pancreatic surgery

Exclusion Criteria:

* Pregnant or lactating females
* Any other major illness or condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in this study
* Subjects who are not a candidate for pancreatic surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lisa States, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] States LJ, Davis JC, Hamel SM, Becker SA, Zhuang H. 18F-6-Fluoro-l-Dopa PET/CT Imaging of Congenital Hyperinsulinism. J Nucl Med. 2021 Jul;62(Suppl 2):51S-56S. doi: 10.2967/jnumed.120.246033. PMID 34230074
- [Background] Palmaz JC. New advances in endovascular technology. Tex Heart Inst J. 1997;24(3):156-9. PMID 9339501
- [Background] Breitwieser W, Price C, Schuster T. Identification of a gene encoding a novel zinc finger protein in Saccharomyces cerevisiae. Yeast. 1993 May;9(5):551-6. doi: 10.1002/yea.320090512. PMID 8322518
- [Background] States LJ, Saade-Lemus S, De Leon DD. 18-F-L 3,4-Dihydroxyphenylalanine PET/Computed Tomography in the Management of Congenital Hyperinsulinism. PET Clin. 2020 Jul;15(3):349-359. doi: 10.1016/j.cpet.2020.03.004. PMID 32498990
- [Background] Shapiro E. The first textbook of electrocardiography. Thomas Lewis: Clinical Electrocardiography. J Am Coll Cardiol. 1983 Apr;1(4):1160-1. doi: 10.1016/s0735-1097(83)80120-x. No abstract available. PMID 6339589
- See also: Study description on CHOP research website — https://www.chop.edu/research-studies/18f-dopa-petct-scan-hyperinsulinism
- See also: CHOP HI Center program webpage — https://www.chop.edu/centers-programs/congenital-hyperinsulinism-center